CLINICAL TRIAL: NCT04334759
Title: DREAM3R: DuRvalumab (MEDI4736) With chEmotherapy as First Line treAtment in Advanced Pleural Mesothelioma - A Phase 3 Randomised Trial
Brief Title: DuRvalumab With chEmotherapy as First Line treAtment in Advanced Pleural Mesothelioma
Acronym: DREAM3R
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: PrECOG, LLC. (Other)
Collaborators: AstraZeneca (Industry); Thoracic Oncology Group Australasia (TOGA) (Unknown); University of Sydney (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DREAM3R; PrE0506 (Other: PrECOG, LLC); TOGA 18/001 (Other: Thoracic Oncology Group Australasia); CTC 0231 (Other: NHMRC Clinical Trials Centre, University of Sydney)
Record Dates: First submitted 2020-04-02; First posted 2020-04-06 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Mesothelioma; Pleural Mesothelioma; Malignant Pleural Mesothelioma
Keywords: Unresectable Mesothelioma; Durvalumab; Anti-Programmed Death-Ligand 1 Antibody; Immune Checkpoint Inhibitor; Ipilimumab; Nivolumab
MeSH Terms: conditions — Mesothelioma; Mesothelioma, Malignant | interventions — durvalumab; Cisplatin; Carboplatin; Pemetrexed; Ipilimumab; Nivolumab

STUDY DESIGN:
Intervention Model Description: First-line chemotherapy with cisplatin or carboplatin and pemetrexed + durvalumab OR physician's choice of either first-line chemotherapy alone, or ipilimumab and nivolumab.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Experimental Arm: Durvalumab + Chemotherapy, then Durvalumab Maintenance (Experimental): Durvalumab + Standard Chemotherapy for 4 to 6 cycles, followed by Maintenance with Durvalumab
  Interventions: Drug: Durvalumab
- Control Arm: Chemotherapy, then Observation (Active Comparator): Standard Chemotherapy for 4 to 6 cycles, followed by Observation
  Interventions: Drug: Standard Chemotherapy
- Control Arm: Ipilimumab and Nivolumab (Active Comparator): Ipilimumab every 6 weeks and Nivolumab every 2 or 3 weeks for up to 2 years.
  Interventions: Drug: Ipilimumab and Nivolumab

INTERVENTIONS:
Drug: Durvalumab — Durvalumab 1500 milligrams (mg) intravenous (IV) every 3 weeks + Cisplatin 75 mg/m² or Carboplatin AUC 5 IV every 3 weeks + Pemetrexed 500 mg/m² IV every 3 weeks for 4 to 6 cycles, followed by maintenance with Durvalumab 1500 mg IV every 4 weeks
  Other Names: MEDI4736; Imfinzi
  Arms: Experimental Arm: Durvalumab + Chemotherapy, then Durvalumab Maintenance
Drug: Standard Chemotherapy — Cisplatin 75 mg/m² or Carboplatin AUC 5 IV every 3 weeks + Pemetrexed 500 mg/m² IV every 3 weeks) for 4 to 6 cycles, followed by Observation
  Other Names: Cisplatin or Carboplatin and Pemetrexed
  Arms: Control Arm: Chemotherapy, then Observation
Drug: Ipilimumab and Nivolumab — Ipilimumab 1 mg/kg every 6 weeks and Nivolumab 360 mg every 3 weeks or 3 mg/kg every 2 weeks for up to 2 years
  Other Names: Yervoy, Opdivo
  Arms: Control Arm: Ipilimumab and Nivolumab

SUMMARY:
Patients with pleural mesothelioma (PM) that cannot be surgically removed will receive standard chemotherapy (cisplatin or carboplatin and pemetrexed) given with durvalumab, a type of immunotherapy, or a treatment chosen by the study doctor, which is either standard chemotherapy or immunotherapy combination (ipilimumab and nivolumab).

Durvalumab is an antibody (a type of human protein) that works by blocking a body substance called Programmed Death-Ligand 1 (PD-L1). Blocking PD-L1 helps the body's immune system attack cancer cells. Research has shown that durvalumab can slow tumor growth and shrink tumors in some people with cancer. Previous studies of combining durvalumab and chemotherapy showed that this combination is active in advanced mesothelioma.

The purpose of this study is to see whether adding durvalumab to standard chemotherapy will improve overall survival (OS) in patients with PM.

DETAILED DESCRIPTION:
Mesothelioma is a malignant tumor of the mesothelial surfaces primarily arising in the thoracic pleura. In the United Kingdom and USA the expected number of cases in the next few decades are 65,000 and 85,000, respectively. Once diagnosed, this disease is rarely cured with a median survival of less than a year.

This is an International, Open-Label, Multi-center, Phase III study. Patients will be randomized 1:1 to receive (a) chemotherapy given with durvalumab versus (b) physician's choice of either chemotherapy alone, or ipilimumab and nivolumab.

Experimental Arm:

- Durvalumab every 3 weeks + standard chemotherapy (cisplatin or carboplatin every 3 weeks + pemetrexed every 3 weeks) for 4 to 6 cycles, followed by durvalumab every 4 weeks until disease progression, unacceptable toxicity or patient withdrawal.

Control Arm: Physician Choice

* Standard chemotherapy (cisplatin or carboplatin every 3 weeks + pemetrexed every 3 weeks) for 4 to 6 cycles followed by observation
* Ipilimumab every 6 weeks and nivolumab every 2 or 3 weeks [physician discretion] for up to 2 years until disease progression, unacceptable toxicity or patient withdrawal .

Tumor assessments and Quality of Life (QOL) forms will be performed at baseline, then at weeks 6, 12, 18, 26, 34, 42, 50 and then every 12 weeks until disease progression. The QOL forms will also be repeated during the first visit after progression.

Mandatory pre-treatment tumor tissue sample (i.e., obtained during a previous procedure or biopsy) for research will also be required. Blood samples for research at 3 time points will be done.

The study is being led jointly by PrECOG as the US sponsor and University of Sydney as the international sponsor.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 years or over) with a histological diagnosis of epithelioid pleural mesothelioma that is not amenable to curative surgical resection. Histological diagnosis requires tumour tissue from an open biopsy, or a core biopsy with a needle of 19 gauge or wider.
* Measurable disease as per modified RECIST 1.1 (mRECIST 1.1) criteria for assessment of response in pleural mesothelioma, without prior radiotherapy to these sites.
* Body weight >30 kg,
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Tumour tissue (Formalin-Fixed Paraffin-Embedded [FFPE]) available from standard of care diagnostic biopsy for PD-L1 testing and other correlative biomarker testing at a central laboratory.
* Life expectancy of at least 12 weeks.
* Adequate blood tests (done within 14 days prior to randomisation) and with values within the ranges specified below. Blood transfusions are permissible if completed at least 7 days prior to treatment start.

  * Haemoglobin ≥ 9.0 g/L
  * Absolute neutrophil count ≥ 1.5 x 10^9/L
  * Platelets ≥ 100 x 10^9/L
  * Total bilirubin ≤ 1.5 x upper limit of normal (ULN) (except participants with Gilbert's Syndrome, who are eligible with bilirubin ≤ 2.5 ULN)
  * Alanine transaminase ≤ 2.5 x upper limit of normal (ULN), unless liver metastases or invasion are present, in which case it must be ≤ 5 x ULN
  * Aspartate aminotransferase ≤ 2.5 x ULN, unless liver metastases or invasion are present, in which case it must be ≤ 5 x ULN
  * Creatinine clearance (CrCl) ≥ 45 mL/min (Cockcroft-Gault formula). NOTE: Carboplatin AUC 5 must be the initial platinum agent of choice in patients with creatinine Cl <60 mL/min but ≥ 45 mL/min, or those with clinically reported hearing loss.
* Patient consent must be appropriately obtained in accordance with applicable local and regulatory requirements. Each patient or legal representative must sign a consent form prior to enrolment in the trial to document their willingness to participate.
* Willing and able to comply with all study requirements, including treatment, timing and/or nature of required assessments.
* Women of childbearing potential must use a reliable means of contraception during treatment and for at least 90 days thereafter. Breastfeeding is not permissible during or for at least 90 days after the final study treatment. Men must have been surgically sterilised or use a barrier method of contraception if they are sexually active with a woman of child bearing potential.
* Evidence of post-menopausal status or negative serum pregnancy test for female pre-menopausal patients. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause.

Exclusion Criteria:

* Non-epithelioid histology (biphasic or sarcomatoid).
* Prior chemotherapy or other systemic anti-cancer or immunotherapy for PM.
* Diagnosis based only on cytology or aspiration biopsy with a needle narrower than 19 gauge.
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g. colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc.]). The following are exceptions to this criterion:

  1. Patients with vitiligo or alopecia
  2. Patients with hypothyroidism (e.g. following Hashimoto syndrome) stable on hormone replacement
  3. Any chronic skin condition that does not require systemic therapy
  4. Patients without active disease in the last 5 years may be included
  5. Patients with celiac disease controlled by diet alone
* Any condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone or equivalent dose of an alternative corticosteroid) or other immunosuppressive medications within 28 days of durvalumab or ipilimumab or nivolumab administration. Intranasal, inhaled or topical steroids or local steroid injections (e.g. intra-articular injection) are permitted in the absence of active autoimmune disease. Standard steroid premedication given prior to chemotherapy or as prophylaxis for imaging contrast allergy should not be counted for this criterion.
* Participants with symptomatic or uncontrolled brain metastases or leptomeningeal disease are excluded.
* Prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T cell co-stimulation or immune checkpoint pathways.
* Current treatment or treatment within the last 12 months with any investigational anti-cancer products.
* Concurrent enrolment in another clinical study testing an anticancer treatment.
* Mean QT interval corrected for heart rate using Fridericia's formula (QTcF) ≥ 470 msec in screening ECG measured using standard institutional method or history of familial long QT syndrome.
* Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of study treatment on protocol. Note: Local surgery of isolated lesions for palliative intent is acceptable. Limited pleural biopsy procedures do not apply.
* No other malignancy that requires active treatment. Participants with a past history of adequately treated carcinoma in situ, non-melanoma skin cancer or lentigo maligna without evidence of disease or superficial transitional cell carcinoma of the bladder are eligible.
* Hearing loss or peripheral neuropathy considered by the investigators to contraindicate administration of either cisplatin, carboplatin or pemetrexed.
* History of allergy or hypersensitivity to investigational product, cisplatin, carboplatin, pemetrexed, ipilimumab, nivolumab or any excipient.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive cardiac failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, active peptic ulcer disease or gastritis, serious chronic gastrointestinal conditions associated with diarrhoea, active bleeding diatheses.
* Hepatitis B, hepatitis C or human immunodeficiency virus (HIV). Exceptions include past or resolved Hepatitis B (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) and patients positive for hepatitis C (HCV) antibody if polymerase chain reaction is negative for HCV RNA. HIV testing is not required in absence of clinical suspicion of HIV.
* Known history of primary immunodeficiency, allogeneic organ transplant, pneumonitis or active tuberculosis.
* Receipt of live attenuated vaccination within 30 days prior to enrolment or within 30 days of receiving durvalumab, ipilimumab, nivolumab.
* Specific comorbidities or conditions or concomitant medications which may interact with the investigational product(s).
* Any condition that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of patient safety or study results.
* Serious medical or psychiatric conditions or social situation that might limit compliance with study requirements, substantially increase risk of incurring adverse events or compromise the ability of the patient to give written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2021-02-18 (Actual); Primary Completion 2025-06-20 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Effects on Overall Survival | Minimum follow-up is 24 months after randomisation.
  Defined as the time from randomisation to the date of death due to any cause.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | Performed at baseline, then at weeks 6, 12, 18, 26, 34, 42, 50 and then every 12 weeks until disease progression (minimum follow-up is 24 months after randomisation).
  Defined as the interval from date of randomisation to the date of first evidence of disease progression or death, whichever occurs first.
Objective Tumour Response Rate (OTRR) | Performed at baseline, then at weeks 6, 12, 18, 26, 34, 42, 50 and then every 12 weeks until disease progression (minimum follow-up is 24 months after randomisation).
  Percentage of participants with either Complete Response (CR) or Partial Response (PR) assessed according to modified Response Criteria in Solid Tumors (RECIST) 1.1 for response in malignant pleural mesothelioma.
Classify and grade participants adverse events as assessed by CTCAE V5.0 | 90 days after last dose of immunotherapy or 30 days after last dose of chemotherapy, whichever is longer.
  Classify and grade participants abnormal laboratory values and/or adverse events.
Health-Related Quality of Life (QOL): QLQ-C30 | Performed at baseline, then at weeks 6, 12, 18, 26, 34, 42, 50, then every 12 weeks until disease progression and at first progression visit (minimum follow-up is 24 months after randomisation).
  European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ-C30), Importance of QOL issues assessed using a four-point scale (1 = not at all, 4 = very much).
Health-Related QOL: LC29 | Performed at baseline, then at weeks 6, 12, 18, 26, 34, 42, 50, then every 12 weeks until disease progression and at first progression visit (minimum follow-up is 24 months after randomisation).
  EORTC Quality of Life Lung Cancer Module (QLQ-LC29), Importance of QOL issues assessed using a four-point scale (1 = not at all, 4 = very much).
Health-Related QOL: EQ-5D-5L | Performed at baseline, then at weeks 6, 12, 18, 26, 34, 42, 50, then every 12 weeks and at first progression visit until disease progression (minimum follow-up is 24 months after randomisation).
  Euro-Quality of Life (EuroQoL) 5 dimension 5 level (EQ-5D-5L) questionnaire, comprising of 5 questions with a score from 1 (no problem) to 5 (extreme problem) and a visual analog scale from 0 (worst) to 100 (best).
Health Care Usage Costs: Hospitalization | Minimum follow-up is 24 months after randomisation.
  Australian Sites Only: Hospitalization costs calculated by applying Australian unit costs to Australian Refined Diagnostic Related Groups (AR DRG) costs for hospitalizations.
Health Care Usage Costs: Scheduled Visits to Health Professionals | Minimum follow-up is 24 months after randomisation.
  Australian Sites Only: Scheduled costs for visits to health professionals collected via Medical Benefits Schedule (MBS).
Health Care Usage Costs: Medications | Minimum follow-up is 24 months after randomisation.
  Australian Sites Only: Scheduled costs for medications collected via the Pharmaceutical Benefits Schedule (PBS).

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Forde, MD, Study Chair — Johns Hopkins University; Anna Nowak, MD, Study Chair — Faculty of Health and Medical Sciences University of Western Australia
Locations (57):
- United States (25):
  - University of California San Diego, La Jolla, California
  - University of Miami, Miami, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - NorthShore University Health System/Kellogg Cancer Center, Evanston, Illinois
  - Johns Hopkins Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Massaschusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Morristown Medical/Atlantic Health, Morristown, New Jersey
  - Jersey Shore University Medical Center, Neptune City, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Memorial Sloan Kettering, New York, New York
  - University of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - Penn State Cancer Institute, Hershey, Pennsylvania
  - Abramson Cancer Cener at Penn Presbyterian Medical Center, Philadelphia, Pennsylvania
  - Allegheny Cancer Center, Pittsburgh, Pennsylvania
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - University of Virginia, Charlottesville, Virginia
- Australia (31):
  - Canberra Hospital, Garran, Australian Capital Territory
  - Blacktown Hospital, Blacktown, New South Wales
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - Coffs Harbour Health Campus, Coffs Harbour, New South Wales
  - Gosford Hospital, Gosford, New South Wales
  - Wyong Hospital, Hamlyn Terrace, New South Wales
  - Nepean Hospital, Kingswood, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - Orange Health Service, Orange, New South Wales
  - Northern Cancer Institute (GenesisCare), Saint Leonards, New South Wales
  - Calvary Mater Newcastle, Waratah, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Icon Cancer Care Wesley, Auchenflower, Queensland
  - Sunshine Coast University Hospital, Birtinya, Queensland
  - Icon Cancer Care Chermside, Chermside, Queensland
  - The Prince Charles Hospital, Chermside, Queensland
  - Townsville University Hospital, Douglas, Queensland
  - Icon Cancer Care South Brisbane, South Brisbane, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Flinders Medical Centre, Bedford Park, South Australia
  - The Queen Elizabeth Hospital, Woodville South, South Australia
  - Royal Hobart Hospital, Hobart, Tasmania
  - Launceston General Hospital, Launceston, Tasmania
  - Monash Health, Clayton, Victoria
  - Peninsula & South Eastern Haematology and Oncology Group, Frankston, Victoria
  - Austin Hospital, Heidelberg, Victoria
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Epworth HealthCare - Richmond, Richmond, Victoria
  - Sunshine Hospital (Western Health), Saint Albans, Victoria
  - Goulburn Valley Health, Shepparton, Victoria
  - Sir Charles Gairdner Hospital (SCGH), Nedlands, Western Australia
- Auckland City Hospital, Grafton, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: No
Data is proprietary

REFERENCES:
- [Background] Kok PS, Forde PM, Hughes B, Sun Z, Brown C, Ramalingam S, Cook A, Lesterhuis WJ, Yip S, O'Byrne K, Pavlakis N, Brahmer J, Anagnostou V, Ford K, Fitzpatrick K, Bricker A, Cummins MM, Stockler M, Nowak AK; Thoracic Oncology Group of Australasia (TOGA) and PrECOG, USA. Protocol of DREAM3R: DuRvalumab with chEmotherapy as first-line treAtment in advanced pleural Mesothelioma-a phase 3 randomised trial. BMJ Open. 2022 Jan 25;12(1):e057663. doi: 10.1136/bmjopen-2021-057663. PMID 35078853
- [Derived] Kindler HL. Understanding the new therapeutic options for mesothelioma. Lancet Oncol. 2021 Oct;22(10):1353-1355. doi: 10.1016/S1470-2045(21)00520-9. Epub 2021 Sep 6. No abstract available. PMID 34499875
- [Derived] Uprety D. CheckMate 743: A Glimmer of Hope for Malignant Pleural Mesothelioma. Clin Lung Cancer. 2021 Mar;22(2):71-73. doi: 10.1016/j.cllc.2020.11.009. Epub 2020 Dec 2. No abstract available. PMID 33358660